CLINICAL TRIAL: NCT04242745
Title: The Effect of an Audible Alarm on the Fluid Consumption of The Elderly Living in a Nursing Home: A Randomized, Controlled Trial
Brief Title: The Effect of Audible Alarm on the Fluid Consumption of the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Perihan ÇETİN, Assistant Professor, PhD,, Izmir Katip Celebi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-7.1/36; 27.07.2017
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: The Elderly
Keywords: Elderly; fluid consumption; fluid deficiency; nursing home; audible alarm
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Procedure/Surgery:The intervention group was given education and a wristwatch which gave an audible alarm to remind them to drink liquid.
  Interventions: Behavioral: Intervention group; Behavioral: Control group
- Control group (No Intervention): The control group was given only education.

INTERVENTIONS:
Behavioral: Intervention group — The elderly in this group were trained using the "For Your Health For Fluid" training booklet and a projection device, and after training, all individuals were given a training booklet. The training was carried out individually in a room reserved for training and took an average of 25-30 minutes.
  A Beyid wristwatch was used. This spoke the time in Turkish, every hour on the hour. In this way, the old people were reminded to drink a glass of liquid each hour. The watch had an alarm capability, and could be taken on to sleep mode at night in order not to wake the old people.
  Arms: Intervention group
Behavioral: Control group — The elderly in this group were trained using the "For Your Health For Fluid" training booklet and a projection device, and after training, all individuals were given a training booklet. The training was carried out individually in a room reserved for training and took an average of 25-30 minutes.
  Arms: Intervention group

SUMMARY:
Research shows that older people need reminders to increase fluid consumption. The aim of the research was to investigate the effect of an audible alarm on the fluid consumption of old people living in a nursing home. The research was conducted as a single-blind, randomized controlled, prospective experimental study on the pre-test post-test model.

The study was performed between 27 July 2017 and 1 February 2018 at a nursing home in the west of Turkey. Out of 979 in nursing home who conformed to the inclusion criteria of the study, 100 (intervention group (n: 50) and control group (n: 50) were voluntarily included in the sample. The intervention group was given education and a wristwatch which gave an audible alarm to remind them to drink liquid, the control group was given only education. The old people in both groups were monitored before the education, after the education, after the audible alarm and 15 days after the audible alarm every three days on total of 12 days. The amount of liquid that the elderly should drink daily was determined according to Gaspar formula.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion in the study were being aged 65 or over, not having a fluid deficiency and living in nursing home.

Exclusion Criteria:

* Exclusion criteria were having an education level of less than primary education
* Being visually or aurally impaired,
* Being bedridden,
* Not being able to take liquids orally, Having health problems such as fever,
* Vomiting, diarrhea or kidney disease causing fluid loss,
* Taking diuretic medication and using more than more than five doses per day,
* Having a diagnosis of a disease such as kidney failure or cardiac insufficiency requiring restriction of fluids, or having a diagnosis of neurological or psychiatric dysfunction, or dementia or Alzheimer's.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Stratified randomization scheme of the intervention and control group is shown below Variable intervention group Control group Total
  Age 65-74 Years 13 13 26 75-84 Years 29 28 57 85 Years and Over 8 9 17 Gender Women 31 30 61 Male 19 20 39 Education Status Primary School 17 18 35 High School and above 33 32 65 Total 50 50 100
Enrollment: 100 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Total amount of fluids taken by the elderly | Through study completion, about three years
  The elderly in the intervention and control groups; before the education (on the 2nd, 3rd and 4th days of the study), after the education (on the 6th, 7th and 8th days of the research), after the audible stimulus (on the 9th, 10th and 11th days of the research), and 15 days after the audible stimulus monitoring (26, On the 27th and 28th days), the total amount of fluid he consumed daily was measured and recorded by the nurse.
Fluid deficit of the elderly | Through study completion, about three years
  The elderly in the intervention and control groups; before the training (on the 2nd, 3rd and 4th days of the study), after the training (on the 6th, 7th and 8th days of the research), after the audible stimulus (on the 9th, 10th and 11th days of the research), and 15 days after the audible stimulus monitoring (26, On the 27th and 28th days), the 24-hour amount of urine and the urine concentration was measured and recorded by the nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Perihan ÇETİN, Assistant Professor, PhD, Study Chair — Izmir Katip Celebi University; İsmet EŞER, Professor, Study Director — Ege University
Locations (1):
- İzmir Katip Çelebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No